CLINICAL TRIAL: NCT03484728
Title: The Interaction Between Conditioned Pain Modulation and Expectation in Understanding the Placebo Effect of Pain Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 574-17_RMB_CTIL
Record Dates: First submitted 2018-01-31; First posted 2018-04-02 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Healthy
Keywords: Conditional pain modulation; pain; placebo
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: CPM was tested before and after the placebo manipulation (body cream application on forearm); based on the expectation of the cream analgesic response (high or low), two types of placebo manipulations were performed for each participant.
Who Masked: Participant, Investigator
Masking Description: The participants were told that the cream has poweful analgetic effect in one session; and that the cream has minmal analgesic effect in another session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-expectation placebo manipulation (Placebo Comparator): application of nonactive body cream on forearm for 10 minutes
  Interventions: Behavioral: placebo manipulation
- Low-expectation placebo manipulation (Other): application of nonactive body cream on forearm for 10 minutes
  Interventions: Behavioral: placebo manipulation

INTERVENTIONS:
Behavioral: placebo manipulation — application of nonactive body cream on forearm

SUMMARY:
The interaction between conditioned pain modulation and expectation in understanding the placebo effect of pain reduction

DETAILED DESCRIPTION:
Conditioned pain modulation (CPM) has recently been coined for the psychophysical protocols that assess the functioning of descending pain inhibitory pathways in humans. There is a growing body of evidence points to the important role of spinal serotonin (5-HT) and noradrenaline (NA) in mediation of pain inhibition via CPM. On the other hand, there is also evidence on synergistic modulatory effect of the opioidergic control on CPM, however this issue is under debates. It seems therefore, that pre-treatment CPM assessment may be relevant for prediction of analgesic drug interaction and additive effects.

Placebo effects are inherent to every treatment and significantly contribute to clinical outcomes even in the presence of strong verum analgesic effects. From a psychological point of view, a series of recent studies supported the nature of the placebo effect as a learning phenomenon wherein verbally-induced expectations, cued and contextual conditioning or social learning are considered as the core mechanisms to produce a benefit. Placebo analgesic effects can be elicited by verbal instructions that generate anticipation for a benefit, thus creating expectations of analgesia. The effect of placebo is, primarily mediated by mu-receptors associated opioidergic neurotransmission. Alike brain structures activated by placebo manipulations, prefrontal cortex, cingulate cortex, PAG and RVM are the most important brain structures involved in initiating of opioid-mediated anti-nociception.

An interesting question that emerges is the extent of overlap between the serotono-noradrenergic analgesia represented by CPM, and opioidergic analgesia represented by expectation-based placebo manipulation, for pain reduction. It seems that the final pathway for the two systems is the descending analgesia tract(s). It is unclear, though, if such final common pathway dictates a limited analgesic effect, i.e., it can only be activated to a certain extent, regardless of which system activates it, and therefore additive effects of expectation and CPM are limited to a certain ceiling. Alternatively, different tracts of descending pain inhibition are activated by each system, and the analgesic effect is additive.

Cognitive cortical brain potentials (especially, a P300 waveform) evoked in response to a combination of rare and frequent innocuous sensory stimuli represent a neurophysiological tool for assessment attention. As this test bases on uncertainty and the expectation of upcoming stimuli, the recording of P300 may be relevant for evaluation cognitive processes associated with expectation-related placebo analgesia.

The main aim of this study is to explore the interaction between serotono-noradrenergic and opioidergic systems of analgesia in healthy subjects. More specifically, the investigator will study whether these two systems work in an additive or a complementary way, and whether the neurophysiological assessment of individual expectation capabilities can predict the placebo magnitude.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Exclusion Criteria:

* attention deficit.
* pain disorders.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change in pain perception | up to 2 weeks
  pain units on a scale of 0-100. 0 no pain. 100 = the maximum pain
Change in conditioned pain modulation (CPM) | up to 2 weeks
  change in pain units on a scale of 0-100. 0 no pain. 100 = the maximum pain

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical center, Neurology Department, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No